CLINICAL TRIAL: NCT01523717
Title: Procalcitonin Decrease Over 72 Hours and Outcome in Patients With Severe Sepsis or Septic Shock
Brief Title: Procalcitonin Monitoring Sepsis Study
Acronym: MOSES
Status: Completed | Type: Observational
Sponsor: Brahms AG (Industry)
Responsible Party: Sponsor
Other Study IDs: brahms-moses
Record Dates: First submitted 2012-01-19; First posted 2012-02-01 (Estimated); Last update posted 2015-03-17 (Estimated); Status verified 2015-03

CONDITIONS: Severe Sepsis; Septic Shock
Keywords: procalcitonin; decrease over 72 hours; severe sepsis; septic shock
MeSH Terms: conditions — Sepsis; Shock, Septic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — EDTA plasma and serum samples

SUMMARY:
The purpose of this study is to investigate the relationship between a procalcitonin decrease over 72 hours and outcome in patients who have severe sepsis or septic shock.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (i.e. >18 years of age) diagnosed with severe sepsis or septic shock as defined in Appendix 1, who are already in the ICU or come from the ED, other wards or directly from out of hospital
* Blood sample collection within 12 hours after diagnosis "severe sepsis or septic shock"No prior enrollment into this study
* Written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adult patients with severe sepsis or septic shock in the emergency department, medical floor, ICU
Sampling Method: Probability Sample
Enrollment: 858 (Actual)
Dates: Start 2011-12; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
28 day all cause mortality | within 28 day safter inlclusion
  participants will be followed up for 28 days

SECONDARY OUTCOMES:
all-cause in-hospital mortality | mortality during hospital stay
  count all death through out stay in the hospital

CONTACTS AND LOCATIONS:
Overall Officials: Nathan Shapiro, MD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (13):
- United States (13):
  - University of California Davis Health System, Sacramento, California
  - Northwestern University, Chicago, Illinois
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Saint Vincent Hospital, Worcester, Massachusetts
  - Detroit Receiving Hospital, Detroit, Michigan
  - Sinai Grace Hospital, Detroit, Michigan
  - Henry Ford Health System, Detroit, Michigan
  - University of Mississippi Medical Center, Jackson, Mississippi
  - New York Methodist Hospital, New York, New York
  - Stony Brook University, New York, New York
  - Carolinas Medical Center, Charlotte, North Carolina
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee